CLINICAL TRIAL: NCT04216134
Title: A Phase I Study of 68GA-PSMA-11 PET Imaging for Biochemically Recurrent Prostate Cancer
Brief Title: 68Ga-PSMA-11 PET for the Diagnosis of Biochemically Recurrent Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 19517; NCI-2019-08625 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 19517 (Other: City of Hope Comprehensive Cancer Center); P30CA033572 (NIH)
Record Dates: First submitted 2019-12-30; First posted 2020-01-02 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Biochemically Recurrent Prostate Carcinoma
MeSH Terms: interventions — gallium 68 PSMA-11; 68Ga-DKFZ-PSMA-11; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Diagnostic (68GA-PSMA-11 PET) (Experimental): Patients receive gallium Ga 68-labeled PSMA-11 IV over less than 1 minute, and then undergo PET over 60 minutes.
  Interventions: Drug: Gallium Ga 68-labeled PSMA-11; Procedure: Positron Emission Tomography

INTERVENTIONS:
Drug: Gallium Ga 68-labeled PSMA-11 — Given IV
  Other Names: (68)Ga labeled Glu-NH-CO-NH-Lys(Ahx)-HBED-CC; (68)Ga-labeled Glu-urea-Lys(Ahx)-HBED-CC; (68)Ga-PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; (68)Gallium-PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; (68Ga)Glu-urea-Lys(Ahx)-HBED-CC; 68Ga-DKFZ-PSMA-11; 68Ga-HBED-CC-PSMA; 68Ga-labeled Glu-NH-CO-NH-Lys(Ahx)-HBED-CC; 68Ga-PSMA; 68Ga-PSMA-11; 68Ga-PSMA-HBED-CC; [68Ga] Prostate-specific Membrane Antigen 11; [68Ga]GaPSMA-11; Ga PSMA; Ga-68 labeled DKFZ-PSMA-11; Ga-68 labeled PSMA-11; Gallium Ga 68 PSMA-11; Gallium-68 PSMA; Gallium-68 PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; GaPSMA; PSMA-HBED-CC GA-68
Procedure: Positron Emission Tomography — Undergo 68GA-PSMA-11 PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging

SUMMARY:
This phase I trial studies the side effects of 68GA-PSMA-11 PET imaging in patients with prostate cancer that has come back (recurrent). Gallium (68Ga) is a radiotracer that binds to a molecule, PSMA, that is found in abundance on most prostate cancer cells. PSMA is short for 'prostate specific membrane antigen'. Diagnostic procedures, such as 68GA-PSMA-11 PET imaging, may help measure a patient's response to earlier treatment, and may help plan the best treatment for prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To provide clinical access to and assess the safety of the investigational agent Gallium Ga 68-labeled prostate specific membrane antigen (PSMA)-11 (68Ga-PSMA-11) positron emission tomography (PET) at City of Hope National Medical Center for patients co-enrolled on Institutional Review Board (IRB) 18517 treatment trial.

OUTLINE:

Patients receive gallium Ga 68-labeled PSMA-11 intravenously (IV) over less than 1 minute, and then undergo PET over 60 minutes.

After completion of study, patients are followed up at 1-3 days, and then at 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Biochemical recurrent prostate cancer
* Karnofsky performance status of >= 50
* The effects of 68Ga-PSMA-11 on the developing fetus are unknown. For this reason, subjects must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for six months following duration of study participation when having sex with a pregnant female or with a female partner of childbearing potential
* Co-enrollment on IRB 18517
* Documented informed consent of the patient. All subjects must have the ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

* Patients should not have any uncontrolled illness including ongoing or active infection
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to 68Ga-PSMA-11
* Use of another concomitant investigational therapy (with the exception of the investigational treatment given in IRB 18517) for prostate cancer within 7 days of scheduled 68Ga-PSMA-11 PET scan
* Unable to tolerate PET scan (i.e. if the patient is claustrophobic or unable to lie still for 30-60 minutes)
* Subjects, who in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-12-12 (Actual); Primary Completion 2022-12-09 (Actual); Study Completion 2022-12-09 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 3 months
  Will be assessed by Common Terminology Criteria for Adverse Events version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Parayno, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States